CLINICAL TRIAL: NCT00963625
Title: Comparison of Transfers of Fresh and Thawed Embryos in Normal Responder Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fertility Center of Las Vegas (Industry)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Bruce Shapiro, M.D., Ph.D., Fertility Center of Las Vegas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAIRB 07-0014
Record Dates: First submitted 2009-08-19; First posted 2009-08-21 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Infertility
Keywords: Blastocyst transfer; endometrial receptivity; IVF; in vitro fertilization; embryo cryopreservation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blastocyst transfer in PTEC cycle (Experimental): Transfer of two blastocysts derived from thawed bipronuclear oocytes that were subject to post-thaw extended culture (PTEC).
  Interventions: Procedure: Embryo cryopreservation
- Fresh blastocyst transfer. (Active Comparator): Transfer of two fresh autologous blastocysts following controlled ovarian stimulation.
  Interventions: Procedure: Fresh blastocyst transfer

INTERVENTIONS:
Procedure: Embryo cryopreservation — Cohort cryopreserved as bipronuclear (2pn) oocytes, then thawed and cultured to the blastocyst stage before transfer to the uterus.
  Arms: Blastocyst transfer in PTEC cycle
Procedure: Fresh blastocyst transfer — Fresh blastocyst transfer following cycle of controlled ovarian stimulation.
  Arms: Fresh blastocyst transfer.

SUMMARY:
This study tests the hypothesis that controlled ovarian stimulation impairs endometrial receptivity in normal responders.

DETAILED DESCRIPTION:
The purpose of this study is to determine if blastocyst transfers in cycles of post-thaw extended culture (PTEC) have different efficacy than transfers of fresh blastocysts in patients with expected normal response to ovarian stimulation.

Multiple studies have found altered endometrial histology and gene expression following controlled ovarian stimulation.

PTEC cycles require cryopreservation of the entire 2pn oocyte cohort in the prior cycle. Once thawed, the embryos are cultured to the blastocyst stage before transfer.

In typical cycles using frozen-thawed embryos, many thawed embryos that appear to survive do not actually resume and continue development. PTEC ensures the transfer of embryos that resumed development and continued developing at least to the blastocyst stage (4-5 days post-thaw).

The viability of a blastocyst in a PTEC cycle has been shown to be on par with that of a fresh blastocyst. Therefore, comparing outcomes of blastocyst transfers in PTEC cycles with that in fresh autologous cycles allows the potential endometrial impact of controlled ovarian stimulation to be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female patient 18 to 40 years of age seeking their first IVF treatment.
* Cycle day 3 FSH less than 10.0 IU/l.
* 8 to 15 antral follicles observed on ultrasound.

Exclusion Criteria:

* Failure to follow the protocol.
* Embryo biopsy.
* Any prior IVF cycle(s).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy (fetal heartbeat observed on ultrasound at 7 weeks gestation) | 7 weeks gestation

SECONDARY OUTCOMES:
Ongoing pregnancy at 10 weeks gestation | 10 weeks gestation
Implantation rate (ratio of the number of fetal heart tones to the number of transferred blastocysts) | 7 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Shapiro, M.D., Ph.D., Principal Investigator — Fertility Center of Las Vegas
Locations (1):
- Fertility Center of Las Vegas, Las Vegas, Nevada, United States

REFERENCES:
- [Derived] Zaat T, Zagers M, Mol F, Goddijn M, van Wely M, Mastenbroek S. Fresh versus frozen embryo transfers in assisted reproduction. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD011184. doi: 10.1002/14651858.CD011184.pub3. PMID 33539543
- [Derived] Shapiro BS, Daneshmand ST, Bedient CE, Garner FC. Comparison of birth weights in patients randomly assigned to fresh or frozen-thawed embryo transfer. Fertil Steril. 2016 Aug;106(2):317-21. doi: 10.1016/j.fertnstert.2016.03.049. Epub 2016 Jul 7. PMID 27397626
- [Derived] Shapiro BS, Daneshmand ST, Garner FC, Aguirre M, Hudson C, Thomas S. Evidence of impaired endometrial receptivity after ovarian stimulation for in vitro fertilization: a prospective randomized trial comparing fresh and frozen-thawed embryo transfer in normal responders. Fertil Steril. 2011 Aug;96(2):344-8. doi: 10.1016/j.fertnstert.2011.05.050. Epub 2011 Jul 6. PMID 21737072